CLINICAL TRIAL: NCT01972555
Title: Single-center Randomized Controlled Trial of Cardiac Function After Minimally Invasive Aortic Valve Implantation (CMILE)
Brief Title: Cardiac Function After Minimally Invasive Aortic Valve Implantation
Acronym: CMILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Peter Svenarud, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMILE
Record Dates: First submitted 2013-10-21; First posted 2013-10-30 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Aortic Valve Stenosis; Heart Valve Diseases
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minimally invasive aortic valve replacement (Experimental): Minimally invasive AVR with either ministernotomy or anterior right-sided minithoracotomy will be performed according to current standard of care practices. Transthoracic echocardiography will be performed preoperatively and at day 1, 4, and 40.
  Interventions: Procedure: Minimally invasive aortic valve replacement
- Conventional aortic valve replacement (Active Comparator): Conventional AVR through a standard median sternotomy will be performed according to current standard of care practices. Transthoracic echocardiography will be performed preoperatively and at day 1, 4, and 40.
  Interventions: Procedure: Conventional aortic valve replacement

INTERVENTIONS:
Procedure: Minimally invasive aortic valve replacement
  Arms: Minimally invasive aortic valve replacement
Procedure: Conventional aortic valve replacement
  Arms: Conventional aortic valve replacement

SUMMARY:
This is a single-center, open-label, randomized controlled trial. Patients scheduled for aortic valve replacement (AVR) at Karolinska University Hospital in Stockholm, Sweden will be eligible. Forty patients will be randomly assigned to either minimally invasive (20 patients) or conventional AVR (20 patients). CE-marked and FDA-approved mechanical and bioprosthetic aortic valves (conventional stented or sutureless bioprostheses) will be implanted. Transthoracic echocardiography will be performed before surgery, and at day 1, 4, and 40. Echocardiographic parameters as well as preoperative clinical characteristics and postoperative clinical outcomes will be registered. Routine blood sampling will be performed pre- and postoperatively. All available data will be collected prospectively. Informed consent will be obtained from patients meeting the inclusion criteria before the initiation of any study-specific procedures.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Severe aortic stenosis defined as aortic valve area of less than 1 cm2 or index area of 0.6 cm2/m2 by echocardiography
* Referred for medically indicated aortic valve replacement
* Sinus rhythm
* Provide written informed consent

Exclusion Criteria:

* Left ventricular ejection fraction less than 0.45
* Presence of any coexisting severe valvular disorder
* Previous cardiac surgery
* Urgent or emergent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Tricuspid Annular Peak Systolic Excursion (TAPSE) | Preoperatively and postoperatively at day 4 and 40
Right ventricular fractional area change | Preoperatively and postoperatively at day 4 and 40
Right ventricular dimensions | Preoperatively and postoperatively at day 4 and 40
Pulsed wave tissue Doppler right venricular velocity | Preoperatively and postoperatively at day 4 and 40

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Sartipy, MD, PhD, Study Chair — Department of Cardiothoracic Surgery and Anesthesiology, Karolinska University Hospital; Reidar Winter, MD, PhD, Study Chair — Department of Cardiology, Karolinska University Hospital
Locations (1):
- Department of Cardiothoracic Surgery and Anesthesiology, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Dalen M, Oliveira Da Silva C, Sartipy U, Winter R, Franco-Cereceda A, Barimani J, Back M, Svenarud P. Comparison of right ventricular function after ministernotomy and full sternotomy aortic valve replacement: a randomized study. Interact Cardiovasc Thorac Surg. 2018 May 1;26(5):790-797. doi: 10.1093/icvts/ivx422. PMID 29325064